CLINICAL TRIAL: NCT06157554
Title: The Effect of Breathing Exercises in Addition to Conventional Treatment on Pain, Normal Joint Movement and Quality of Life in Frozen Shoulder Patients: a Randomized Controlled Trial
Brief Title: The Effect of Breathing Exercises in Addition to Conventional Treatment in Frozen Shoulder Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Assistant professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Frozen shoulder
Record Dates: First submitted 2023-11-21; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Frozen Shoulder; Pain; Quality of Life
MeSH Terms: conditions — Bursitis; Pain | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Respiratory exercises will be applied in addition to conventional treatment for frozen shoulder patients.
  Interventions: Other: Breathing Exercises; Other: Conventional treatment
- Control Group (Other): For frozen shoulder patients, 15 conventional treatment programs will be applied.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Breathing Exercises — During the exercise sessions, participants will be seated in a chair. In the first five and last five minutes of the session, they will be instructed to focus on their breathing and the sensations produced in the body while sitting comfortably in a relaxed position with all joints in the chairs with their eyes closed. After the initial 5 minutes of relaxed breathing, participants will be instructed to perform diaphragmatic and costal breathing for 10 minutes. After 5 minutes of diaphragmatic breathing, the patient will be rested for 1 minute and then 5 minutes of costal breathing will be performed. While doing coastal breathing, patients will be asked to place their hands on their costas, take a deep breath and inflate the bottom of their hands; then they will be asked to exhale the breath they take in a longer (1:2) time.
  Arms: Intervention group
Other: Conventional treatment — Ultrasound, hotpack and TENS will be applied to both control and study groups as physical therapy modality. Then 15 sessions of Codman exercises, normal range of motion exercises and stretching exercises will be applied to both groups.

SUMMARY:
The study aimed to investigate the effect of breathing exercises in addition to conventional treatment on pain, normal joint movement and quality of life in patients with frozen shoulder.

A simple random number table will randomly divide participants into two groups. The study group (20 participants) will be given 15 sessions of respiratory exercises in addition to the 15 sessions of physiotherapy provided routinely for treatment. The control group (20 participants) will receive 15 sessions of physiotherapy services in addition to the routine 15 sessions of the physiotherapy department.

DETAILED DESCRIPTION:
After completing the demographic information form, a visual analog scale will be used for pain intensity, a Baseline digital goniometer will be used to measure the normal joint range of the shoulder girdle, and a Short form SF-36 will be used for quality of life. All participants will be evaluated before and after 15 sessions. The same assessments will be performed in both groups. The evaluations are expected to last 40 minutes in total.

The study group (20 participants) will be given 15 sessions of respiratory exercises in addition to the 15 sessions of physiotherapy provided routinely for treatment. The control group (20 participants) will receive 15 sessions of physiotherapy services in addition to the routine 15 sessions of the physiotherapy department.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having a diagnosis of a frozen shoulder,
* Volunteering to participate in the study
* Not having any problem that may prevent respiratory exercise.

Exclusion Criteria:

* Not volunteering to participate in the study,
* Having undergone upper extremity surgery,
* History of previous shoulder surgery, shoulder subluxation or dislocation,
* Any mental or sensory problems,
* Acute infection or chronic disease of neurological, psychiatric, orthopedic, cardiological, rheumatological, etc. origin,
* Having any respiratory disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3 weeks
  In this study, the severity of shoulder pain will be evaluated with the Visual Analogue Scale. According to the VAS, pain intensity is graded as "no pain" 0 points and "worst unbearable pain" 10 points (10 cm scale).
The Short Form-36 Quality of Life Questionnaire | 3 weeks
  The Short Form-36, frequently used to assess quality of life, will be used. SF-36 consists of eight subscales including physical function, physical role, emotional function, social function, general health, mental health, pain and wellness. Each subscale scores between 0-100, and the scale is directly proportional to quality of life. A score of 100 indicates the best health status and a score of 0 indicates the worst health status.
Range of motion | 3 weeks
  In the study, a digital goniometer, which has been validated and reliable, was used to objectively evaluate the normal range of motion of the shoulder. Normal range of motion of the shoulder will be evaluated by measuring the range of motion of shoulder flexion, extension, abduction, internal rotation and external rotation movements.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided